CLINICAL TRIAL: NCT02537743
Title: Open-labeled, Multicenter, Non-interventional, Prospective PRO Registry for Patients With First Line Treatment for Advanced RCC Using a Tablet-technology Based Digital Device
Brief Title: Prospective Patient Reported Outcomes (PRO) Registry in Patients With Advanced Renal Cell Carcinoma
Acronym: PROKidney
Status: Completed | Type: Observational
Sponsor: iOMEDICO AG (Industry)
Responsible Party: Sponsor
Other Study IDs: IOM - 04302
Record Dates: First submitted 2015-08-26; First posted 2015-09-02 (Estimated); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Renal Cell Carcinoma
Keywords: Patient Reported Outcomes
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Evaluation of patient reported outcomes ( PRO) regarding typical ailments in the REAL LIFE Renal Cell Carcinoma population

DETAILED DESCRIPTION:
The PRO Kidney project will recruit a representative cohort of patients with advanced renal cell carcinoma (RCC) treated with systemic antiproliferative therapies such as TKIs, mTOR inhibitors, cytokines, antiVEGF or immune therapy. The aim of this study is to collect data on the effectiveness and patients´quality of life on preference in the real life setting.

Patient Reported Outcomes ( PRO) are assessed by a questionnaire consisting Functional Assessment of Cancer Therapy ( FACT) Kidney Syndrome Index 19 (FKSI 19) completed by four questions assessing ailments about changes in skin of hands/feet, taste, color of hair and mouth scores.

13 Questions about Fatigue assessed with the Functional Assessment of Chronic IIlness Disease.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed renal cell carcinoma
* Start of the first line systemic treatment
* Ability to read and understand German
* Written informed consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with advanced (inoperable or metastatic) renal cell cancer at the start of the first line antitumoral therapy
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2015-08-19 (Actual); Primary Completion 2021-02-19 (Actual); Study Completion 2021-02-19 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Measure (Patient Reported Outcomes (PRO) regarding typical ailments in the real Life RCC population) | 24 months
  Patient Reported Outcomes (PRO) regarding typical ailments in the real Life RCC population

SECONDARY OUTCOMES:
Secondary Outcome Measures (Patient Reported Outcomes (PRO) regarding the impact of treatment on daily life) | 24 months
  Patient Reported Outcomes (PRO) regarding the impact of treatment on daily life

CONTACTS AND LOCATIONS:
Overall Officials: Tilman Kirste, MD, Study Chair — medical practise for oncology
Locations (1):
- Multiple sites all over Germany, Multiple Locations, Germany

IPD SHARING:
Plan to Share IPD: No